CLINICAL TRIAL: NCT01294514
Title: Novel Cardio-Respiratory Parameter in Healthy Volunteers
Brief Title: Novel Non-Invasive Monitoring Parameter in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0132
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-01-10 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: No Conditions; Focus is Respiratory Rate
Keywords: Respiratory Rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy volunteers ASA Class 1

SUMMARY:
The purpose of this study is to study Non-Invasive Performance evaluation of monitoring algorithm.

DETAILED DESCRIPTION:
Assess equivalency, performance, and accuracy of a new monitoring algorithm in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 or older
* Subject is willing and able to provide written consent

Exclusion Criteria:

* Severe contact allergies to standard adhesive materials
* Subjects with abnormalities that may prevent proper application of the device
* Women who are pregnant or lactating
* Subjects with significant Arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Principal Investigator — Medtronic - MITG
Locations (1):
- Covidien- RMS, Boulder, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Respiration Rate in Healthy Volunteers: Healthy volunteer participants were monitored for 30 minute period to collect respiratory rate information from non-invasive sensors.
  Covidien Respiration Rate, Transthoracic Impedance and Overscored Endtidal Carbon Dioxide.
Period: Overall Study
Arm/Group | Respiration Rate in Healthy Volunteers
Started | 27
Completed | 26
Not Completed | 1
Not completed — Excluded due to Arrhythmia | 1

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- Healthy Volunteers: Healthy volunteers were studied
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: The Covidien Nellcor Respiration Rate Software Shall Determine Respiration Rate Measured as Mean and Standard Deviation With Accuracy That is Non-inferior to Predicate Device.
Description: Mean and standard deviations of respiration rates collected from healthy volunteers were compared between Covidien Respiration Rate Software, Transthoracic Impedance and Overscored End-Tidal Carbon Dioxide Waveforms. Each volunteer served as its own control.
Time Frame: Participants were monitorerd on average of 30 minute period
Population: One participant was excluded from the analysis based on cardiac arrhythmia
Measure: Mean (Standard Deviation); unit: Breaths Per Minute (BrPM)
Groups:
- Respiration Rate From Covidien Respiration Rate Software: Respiration Rate determined by novel plethysmographic analysis
- Respiration Rate From Endtidal Carbon Dioxide: Respiration Rate determined by manual overscoring of capnography waveforms.
- Respiration Rate From Transthoracic Impedance: Respiration Rate determined by Transthoracic Impedance
Arm/Group | Respiration Rate From Covidien Respiration Rate Software | Respiration Rate From Endtidal Carbon Dioxide | Respiration Rate From Transthoracic Impedance
Number analyzed (Participants) | 26 | 26 | 26
Breaths Per Minute (BrPM) | 13.2 (3.0) | 13.8 (3.2) | 19.5 (9.4)

2. Secondary Outcome: The Covidien Nellcor Respiration Rate Software Shall Calculate Respiration Rate With a Root Mean Square Difference (RMSD) of < 3 Breaths Per Minute Compared With a End-Tidal Carbon Dioxide Waveforms, With 95% Confidence.
Description: The data used for analysis consisted of multiple simultaneous measures of RR_TTI, RR_V1.0 and RR_EtCO2 for each subject. Given N sets of simultaneous RR values for each of P patients, the simultaneous RR values were used to calculate a pair of RMSD values for each subject.
  The two RMSD values, RMSDRR_V1.0_vs_EtCO2, and RMSDTTI_vs_EtCO2, quantify the mean absolute difference in simultaneous estimates of respiratory rate between RR_V1.0 compared with RR_EtCO2 and RR_TTI compared with RR_EtCO2, respectively for the subjects with 95% confidence of mean ± 3.38 BrPM. The Measure type is Number and represents the RMSD of Covidien Nellcor Respiration Rate Software
Time Frame: Participants were monitored on average of 30 minute periods
Population: One participant was excluded from the data analysis based on cardiac arrhythmia
Measure: Number; unit: Breaths Per Minute (BrPM)
Groups:
- Healthy Volunteers: Covidien Respiration Rate, Transthoracic Impedance and Overscored Endtidal Carbon Dioxide derived respiration rates were recorded on all the volunteers simultaneously.
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 26
Breaths Per Minute (BrPM) | 0.84

3. Post Hoc Outcome: Calculate Covidien Respiration Rate Software Accuracy as Mean Error +/- Standard Deviation
Description: The Covidien Nellcor Respiration Rate Software shall calculate respiration rate as mean error of +/- standard deviation.
Time Frame: Overall average
Population: One participant was excluded from the data analysis based on cardiac arrhythmia
Measure: Mean (Standard Deviation); unit: Breaths Per Minute (BrPM)
Groups:
- Healthy Volunteers: Covidien Respiration Rate, Transthoracic Impedance and Overscored Endtidal Carbon Dioxide.
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 26
Breaths Per Minute (BrPM) | 0.37 (0.78)

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Healthy Volunteers: A selection of subjects from the general population from ages 18 - 50.
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes